CLINICAL TRIAL: NCT04468126
Title: Impact on Mortality of an Oxygenation Strategy Including Standard Oxygen Versus High Flow Nasal Cannula Oxygen Therapy in Patients With Acute Hypoxemic Respiratory Failure: a Prospective, Randomized Controlled Trial.
Brief Title: Standard Oxygen Versus High Flow Nasal Cannula Oxygen Therapy in Patients With Acute Hypoxemic Respiratory Failure
Acronym: SOHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOHO
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure; Hypoxemic Respiratory Failure
Keywords: acute hypoxemic respiratory failure; de novo respiratory failure; high-flow nasal oxygen; standard oxygen
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard oxygen group (Active Comparator): In order to maintain SpO2 between 92 and 96%
  Interventions: Other: Standard oxygen
- high-flow nasal cannula oxygen group (Experimental): At least 50 L/min adjusted in order to maintain SpO2 between 92 and 96 %
  Interventions: Other: High-flow nasal oxygen therapy

INTERVENTIONS:
Other: Standard oxygen — Standard low flow oxygen therapy through facemask or non-rebreathing mask at least 10 L/min.
  Arms: standard oxygen group
Other: High-flow nasal oxygen therapy — Humidified and heated oxygen with a gas flow at least 50 l/min through nasal cannula and inspired fraction of oxygen adjusted in order to maintain a SpO2 between 92 and 96%
  Arms: high-flow nasal cannula oxygen group

SUMMARY:
First-line therapy of patients with acute respiratory failure consists in oxygen delivery through standard oxygen, high-flow nasal oxygen therapy through cannula or non-invasive ventilation. Non-invasive ventilation in acute hypoxemic respiratory failure is not recommended. In a large randomized controlled study, high-flow nasal oxygen has been described as superior to non-invasive ventilation and standard oxygen in terms of mortality but not of intubation. Paradoxically in immunocompromised patients, high-flow nasal oxygen has not been shown to be superior to standard oxygen. To improve the level of evidence of daily clinical practice, we propose comparing high-flow nasal oxygen versus standard oxygen, in terms of mortality in all patients with acute hypoxemic respiratory failure

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients older than 18 years with an acute hypoxemic respiratory failure will be enrolled if they meet all the following criteria:

* Respiratory rate >25 breaths/min whatever the oxygen support
* Pulmonary infiltrate,
* PaO2/FiO2 ≤200 mmHg
* Informed consent from the patient or relatives.

Exclusion Criteria:

* PaCO2 > 45 mm Hg
* Need for emergent intubation: pulse oximetry < 90% with maximum oxygen support, respiratory arrest, cardiac arrest, or Glasgow coma scale below 8 points
* Hemodynamic instability defined by signs of hypoperfusion or use of vasopressors > 0.3 µg/kg/min
* Glasgow coma scale equal to or below 12 points
* Exacerbation of chronic lung disease including chronic obstructive pulmonary disease (grade 3 or 4 of Gold classification), or another chronic lung disease with long term oxygen or ventilatory support
* Cardiogenic pulmonary edema as main reason for acute respiratory failure
* Coronavirus SARS-2 infection as reason for acute respiratory failure (the SOHO-COVID study has been completed)
* Post-extubation respiratory failure within 7 days after extubation,
* Post-operative patients within 7 days after abdominal or cardiothoracic surgery,
* Do not intubate order;
* Already included in the study, refusal to participate or participation in another interventional study with the same primary outcome.
* Patients without any healthcare insurance scheme or not benefiting from it through a third party,
* Persons under law protection, namely minors, pregnant or breastfeeding women, persons deprived of their liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality at 28 days after randomization | Day 28
  Death between randomization and 28 days after randomization

SECONDARY OUTCOMES:
Failure of the oxygenation strategy between randomization and D28 | Day 28
  Intubation between randomization and D28
Mortality in ICU, in hospital, and day 90 | Day 90
  Death between randomization and end of stay in ICU, hospital. Death between randomization and day 90.
Number of ventilation free days at Day 28 | Day 28
  days alive and without intubation between day 1 and day 28
Duration of ICU and hospital stay | Day 90
  ICU and hospital stay between randomisation and end of stay in ICU and hospital
Complications during the ICU stay | Day 90
  Complications during the ICU stay include: septic shock, nosocomial pneumonia, cardiac arrhythmia, and cardiac arrest.
Dyspnea | Hour 1
  feeling is evaluated using a 5-point Likert scale, indicating marked improvement (+2), slight improvement (+1), no change (0), slight deterioration (-1) and marked deterioration (-2)
Comfort | Hour [1;6]
  comfort is evaluated using a 100-mm visual-analogue scale, from 0, i.e. "no discomfort", to100, i.e. "maximal imaginable discomfort"
Level of oxygenation | Hour [1;6]
  Oxygenation is assessed by arterial blood gas sample
Organ Failure during the 48 hours after intubation. | Day 28
  Organ failure is evaluated by the Sepsis-related Organ Failure Assessment (SOFA) score during the 48 hours after intubation.
Duration between the time when prespecified criteria of intubation are met and intubation | Day 28
  interval between the time when prespecified criteria of intubation are met and intubation
Duration between treatment initiation and intubation | Day 28
  Interval between treatment initiation and intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre FRAT, PhD, Principal Investigator — CHU Poitiers
Locations (1):
- CHu Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No
Our institution does not have a data sharing platform.

REFERENCES:
- [Derived] Frat JP, Coudroy R, Quenot JP, Guitton C, Badie J, Gacouin A, Ehrmann S, Demoule A, Jarousseau F, Carteaux G, Rigaud JP, Reignier J, Sedillot N, Contou D, Beloncle F, Daubin C, Dureau AF, Fatah A, Besse MC, Ferre A, Turbil E, Merdji H, Galerneau LM, Lacombe B, Richard JC, Romen A, Delbove A, Prat G, Lautrette A, Colin G, Soum E, Bourdin G, Hernandez G, Ragot S, Thille AW; REVA network. Effect of high-flow nasal cannula oxygen versus standard oxygen on mortality in patients with acute hypoxaemic respiratory failure: protocol for a multicentre, randomised controlled trial (SOHO). BMJ Open. 2024 Oct 23;14(10):e083232. doi: 10.1136/bmjopen-2023-083232. PMID 39448217
- [Derived] Frat JP, Quenot JP, Badie J, Coudroy R, Guitton C, Ehrmann S, Gacouin A, Merdji H, Auchabie J, Daubin C, Dureau AF, Thibault L, Sedillot N, Rigaud JP, Demoule A, Fatah A, Terzi N, Simonin M, Danjou W, Carteaux G, Guesdon C, Pradel G, Besse MC, Reignier J, Beloncle F, La Combe B, Prat G, Nay MA, de Keizer J, Ragot S, Thille AW; SOHO-COVID Study Group and the REVA Network. Effect of High-Flow Nasal Cannula Oxygen vs Standard Oxygen Therapy on Mortality in Patients With Respiratory Failure Due to COVID-19: The SOHO-COVID Randomized Clinical Trial. JAMA. 2022 Sep 27;328(12):1212-1222. doi: 10.1001/jama.2022.15613. PMID 36166027